CLINICAL TRIAL: NCT04074109
Title: Feasibility of At-Home Telehealth Yoga for Treating Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Peter Bayley, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAY0006AGG; R34AT010364 (NIH)
Record Dates: First submitted 2019-08-05; First posted 2019-08-29 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain; Musculoskeletal Pain
Keywords: telehealth; yoga
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: End-of-treatment assessments will be conducted by an assessor who is blind to treatment modality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teleyoga (Experimental): group will receive instruction via computer tablet
  Interventions: Combination Product: Teleyoga
- In-person yoga (Active Comparator): group will receive instruction in-person
  Interventions: Behavioral: In-person yoga

INTERVENTIONS:
Combination Product: Teleyoga — the yoga protocol will be delivered via a tablet computer to groups of participants
  Arms: Teleyoga
Behavioral: In-person yoga — the yoga protocol will be delivered by a yoga instructor in the room to group of participants
  Arms: In-person yoga

SUMMARY:
This feasibility study will evaluate yoga as a treatment for chronic musculoskeletal pain. The experimental treatment is yoga delivered via a tablet computer to participants at home ("teleyoga"). First, the investigators will develop a suitable protocol for teleyoga. Second, the investigators will demonstrate the feasibility of conducting a randomized controlled trial involving randomization to teleyoga or in-person yoga groups.

DETAILED DESCRIPTION:
The first phase of the study is not randomized. In this phase, the first group of participants (n=10) will all participate in a tele-yoga class using an iPad loaned to them by the study. They will attend this treatment session from the comfort of their home or a location of their choice. Yoga treatment will last 12 weeks. At the end of treatment, veterans will provide feedback by completing a satisfaction questionnaire to rate various aspects of the teleyoga (e.g. technical challenges, ability to perform yoga through the video-conferencing platform, problems that occurred, and recommendations to improve the class, etc). The teleyoga protocol will be modified on the basis of this feedback and will be tested on a second group of participants (n=10). The second phase of the study will involve randomization of a further group of participants (n=30) to either the teleyoga developed in phase one, or in-person yoga.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Medical clearance for participation by VA primary care provider
* Diagnosis of musculoskeletal pain > 6 months
* Minimum pain intensity of 4 at screening on 0-10 scale
* Any psychotropic treatments stable for at least 4 weeks before study
* English literacy
* Wireless Internet connection at home

Exclusion Criteria:

* Current participation in another clinical trial
* Back surgery within the last 12 months
* Back pain related to a specific underlying cause, disease, or condition
* Baseline pain <4 or >9 on 0-10 scale
* Unstable, serious coexisting medical illness
* Unstable, serious coexisting mental illness
* Attended or practiced yoga ≥1 time in the past 12 months
* Active current suicidal plan or intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Derived] Mahoney L, Pahade S, Mahoney H, Fitz K, Keaney A, Parker-Bridges K, Francisco JM, Lau A, Hitching R, Walker B, Gupta A, Jo B, Lohnberg JA, Clark JD, Bayley PJ. Randomized Feasibility Trial of Teleyoga versus In-Person Yoga for Treating Chronic Musculoskeletal Pain in Veterans. Res Sq [Preprint]. 2025 Jun 23:rs.3.rs-6265068. doi: 10.21203/rs.3.rs-6265068/v1. PMID 40678237

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Teleyoga | In-person Yoga
Started | 18 | 16
Completed | 13 | 8
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teleyoga | In-person Yoga | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (18.9) | 62 (15.1) | 61.06 (17.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 12 | 12
  Male | 18 | 4 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Multi-Dimensional Treatment Satisfaction Measure
Description: A participant satisfaction measure [score range: 0 to 4]. The higher the value, the greater the treatment satisfaction
Time Frame: after 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teleyoga | In-person Yoga
Number analyzed (Participants) | 13 | 8
score on a scale | 3.2 (0.36) | 3.6 (0.19)
Statistical Analysis 1: Comparison: Teleyoga vs In-person Yoga; Test type: Other — This is a feasibility study which is not powered for efficacy. Therefore no formal statistical tests are used; This is a feasibility study which is not powered for efficacy. Therefore no formal statistical tests are used; This is a feasibility study which is not powered for efficacy. Therefore no formal statistical tests are used
Statistical Analysis 2: Comparison: Teleyoga vs In-person Yoga; This is a feasibility study which is not powered for efficacy. Therefore no formal statistical tests are used. We report percentages and frequencies to show feasibility; Test type: Other; This is a feasibility study which is not powered for efficacy. Therefore no formal statistical tests are used

2. Primary Outcome: Adherence to the Treatment Protocol
Description: % of randomized patients who attend ≥65% of treatment sessions
Time Frame: during 12 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Teleyoga | In-person Yoga
Number analyzed (Participants) | 18 | 16
Participants | 10 | 7

3. Primary Outcome: Attrition
Description: number of randomized patients who drop out of treatment
Time Frame: during 12 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Teleyoga | In-person Yoga
Number analyzed (Participants) | 18 | 16
Participants | 5 | 8

ADVERSE EVENTS:
Time Frame: baseline to end of treatment (12 weeks)
Arm/Group | Teleyoga | In-person Yoga
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

LIMITATIONS AND CAVEATS:
Recruitment and treatment took place during the COVID-19 pandemic which may have influenced the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT04074109/Prot_SAP_ICF_000.pdf